CLINICAL TRIAL: NCT03222063
Title: A Study to Assess the Effectiveness of Play Interventions on Anxiety Among Hospitalized Children in Selected Hospital of Yamuna Nagar, Haryana
Brief Title: Effectiveness of Play Interventions on Anxiety Among Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Pooja saharan, Student, M.Sc. Nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 785
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Anxiety
Keywords: Play interventions, anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental Group:
  Experimental group consists of 30 hospitalized children.In Experimental group after taking pretest on 1st day play interventions were introduced to the children and instructions regarding the way to play with all the interventions were provided to the children. Though all the children were free to choose the play yet the younger children were given simple and easy play interventions such as drawing, coloring etc. to obtain more sensory experience whereas the older children were offered play interventions such as puzzle, building blocks, ludo etc. with high cognitive demand. The play interventions were administered for 1 hour daily for continuous 5 days.Post test assessment of anxiety was done on 5th day.
  Interventions: Other: Play interventions
- Comparison group (No Intervention): Comparison Group: 30 hospitalized children were selected by purposive sampling in comparison group. Pretest anxiety was measured on 1st day . No intervention was administered. only usual medical and nursing care was administered to the hospitalized children. Post test assessment of anxiety was done on 5th day.

INTERVENTIONS:
Other: Play interventions — The following play were included in play interventions i.e building blocks, paint, puzzles, crayons, doctor set, ludo, snake and ladder. All hospitalized children in experimental group received play interventions at bed side. Taking into consideration the busy clinical setting, each participant received continuously 1 hour of hospital play interventions each day for continuous 5 days. Although the hospitalized children were free to choose according to their choice but still the younger children would be engaged in play such as doctor set, Drawing etc. to obtain more sensory experience and older children were offered play interventions such as puzzle, building blocks, ludo etc.with high cognitive demand.
  Arms: Experimental group

SUMMARY:
The study evaluates the effectiveness of play interventions on anxiety among hospitalized children in selected hospital of Yamuna Nagar, Haryana. Quasi experimental approach was adopted. 60 (30 in experimental and 30 in comparison)hospitalized children were selected by purposive sampling technique.Hospitalized children in experimental group were provided play interventions whereas the children in Comparison group received only usual medical and nursing care.

DETAILED DESCRIPTION:
TSetting was selected by randomization (by lottery method) first selected two rooms from General Pediatric Wards were coded as E1 (Experimental 1) and E2 (Experimental 2) whereas next two were coded as C1 (Comparison 1) and C2 (Comparison 2).

From the selected settings 60 subjects (30 in experimental and 30 in Comparison) were selected by purposive sampling technique. Assessment of anxiety (Pre-test) of the hospitalized children admitted in Aashirwad Hospital was done in experimental group and Comparison group on 1st day. In Experimental group after taking pretest play interventions were introduced to the children and instructions regarding the way to play with all the interventions were provided to the children. Though all the children were free to choose the play yet the younger children were given simple and easy play interventions such as drawing, coloring etc. to obtain more sensory experience whereas the older children were offered play interventions such as puzzle, building blocks, ludo etc. with high cognitive demand. The play interventions were administered for 1 hour daily from day 1 to day 5 whereas in Comparison group all the subjects were given usual general nursing and medical care for continuous 5 days. No intervention was administered to the comparison group. Posttest anxiety was assessed on 5th day.

Intervention to the control group was given after the accomplishment of Post test for ethical consideration.

ELIGIBILITY:
Inclusion Criteria:

* The study include hospitalized children who were:

  1. aged 6-12 yrs. admitted in the pediatric general medical unit.
  2. anxious due to hospitalization.
  3. willing to participate in the study.
  4. alert, oriented, comprehend and able to speak and understand Hindi language.

Exclusion Criteria:

The study exclude hospitalized children who were:

* 1. treated as outpatient

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Structured anxiety rating scale | 05 minutes
  It include:
  * Total 30 items and consists of 4 areas that includes apprehension, Nervousness/tension, discomfort and irritability.
  * The maximum score is 90 and minimum 0. The level of anxiety were categorized into 4 categories as shown in table no. 3.3
  Anxiety among hospitalized children was measured by using structured anxiety rating scale which was categorized as no anxiety(0-23), mild to moderate(24-45), severe(46-68) and panic anxiety(69-90).

CONTACTS AND LOCATIONS:
Overall Officials: Ms. Eenu Rani, M.Sc.Nursing, Study Director — Maharishi Markandeshwar University

REFERENCES:
- [Background] Potasz C, De Varela MJ, De Carvalho LC, Do Prado LF, Do Prado GF. Effect of play activities on hospitalized children's stress: a randomized clinical trial. Scand J Occup Ther. 2013 Jan;20(1):71-9. doi: 10.3109/11038128.2012.729087. Epub 2012 Oct 18. PMID 23078405
- [Background] Nabors L, Bartz J, Kichler J, Sievers R, Elkins R, Pangallo J. Play as a mechanism of working through medical trauma for children with medical illnesses and their siblings. Issues Compr Pediatr Nurs. 2013 Sep;36(3):212-24. doi: 10.3109/01460862.2013.812692. Epub 2013 Jul 11. PMID 23845098